CLINICAL TRIAL: NCT01214057
Title: Preliminary Study to Assess the Effects of Total Intravenous Anesthesia With Propofol/Remifentanyl Compared to Sevoflurane/Remifentanyl for Endoscopic Sinus Surgery: Novel Approach.
Brief Title: Total Intravenous Anesthesia (TIVA) vs. Inhaled Anesthesia for Endoscopic Sinus Surgery.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was terminated for patient recruitment difficulty and interim power analysis
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Davide Cattano, Associate Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-10-0014
Record Dates: First submitted 2010-08-04; First posted 2010-10-04 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Chronic Rhinosinusitis
Keywords: chronic rhinosinusitis; endoscopic sinus surgery; TIVA; surgical field visualization
MeSH Terms: interventions — Propofol; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total Intravenous Anesthesia (Experimental): Total Intravenous Anesthesia (TIVA) with propofol and remifentanyl
  Interventions: Drug: Propofol and Remifentanyl
- Inhaled Anesthesia (Active Comparator): Inhaled anesthesia with sevoflurane and remifentanyl.
  Interventions: Drug: Sevoflurane and Remifentanyl

INTERVENTIONS:
Drug: Propofol and Remifentanyl — Anesthesia will be induced with lidocaine 0.5 mg kg, propofol infusion at 250 mcg/kg/min (to reduce visual bias of propofol infusion) and total volume infused will be adjusted for an induction dose of 2-3 mg/kg before bolus of muscle relaxant, rocuronium 0.5 mg kg in both SR and PR groups. Remifentanil infusion will be started at a rate of 0.4 mcg/kg/min 1-2 minutes before the propofol infusion and a 100 ml 0.9% normal saline bag will be used to blind surgeons in the sevoflurane group. The target mean arterial blood pressure (MAP) will be maintained at 70-80 mm Hg by adjusting the propofol concentration within their range (100-150 mg ml for propofol) according to the anaesthesiologist's judgement and by surgeon request. If this failed, the remifentanil rate will be adjusted by 0.05 mg kg min.
  Other Names: Propofol brand name is Diprivan; Remifentanyl brand name is Ultiva
  Arms: Total Intravenous Anesthesia
Drug: Sevoflurane and Remifentanyl — Sevoflurane 1-3% will be administered in group SR, and the infusion of propofol will be stopped. After intubation remifentanil infusion will be changed to 0.2 mcg/kg/min. The target mean arterial blood pressure (MAP) will be maintained at 70-80 mm Hg by adjusting the sevoflurane concentration within their range (between 1-3 vol% for sevoflurane) according to the anaesthesiologist's judgement and by surgeon request.If this failed, the remifentanil rate will be adjusted by 0.05 mg kg min.In order to limit the amount of fluids remifentanil wil be diluted at a concentration of 4 mg in 100 ml.
  Other Names: Remifentanyl brand name is Ultiva; Sevoflurane brand name is Ultane and Sojourn
  Arms: Inhaled Anesthesia

SUMMARY:
The purpose of this study is to compare total intravenous anesthesia to inhaled anesthesia in endoscopic sinus surgery for chronic sinusitis. The investigators will compare bleeding during surgery, duration of surgery, blood flow to the nose and other parameters. The investigators hypothesize that total intravenous anesthesia decreases bleeding and improves the view during surgery.

DETAILED DESCRIPTION:
Endoscopic sinus surgery (ESS) has revolutionized the surgical treatment of chronic sinus disease, permitting outpatient sinus surgery with minimal morbidity. Previously performed using local anesthesia, the majority of patients and surgeons now prefer general anesthesia for comfort, stress containment and relative ease of accomplishing the surgical objectives1.

A critical factor in ESS is the amount of blood in the surgical field. Even for experienced endoscopists, significant bleeding may compromise the safety and completeness of the intended procedure. In addition, increased bleeding requires frequent suctioning therefore decreasing the overall efficiency of the operation and prolonging operative time.

Techniques commonly used to minimize bleeding include but are not limited to topical decongestion, local injection of vasoconstrictors, maintaining normothermia, head elevation, and controlled hypotension. However, controlled hypotension is potentially a source of excessive vasodilatation and risk factor for ischemic events. In fact, a considerable amount of data has shown that the blood pressure and intraoperative bleeding are not necessarily related, and hypotension on its own does not necessarily improve the surgical field2, 3.

In order to maintain a good peripheral perfusion the choice of anesthetics and other drugs is an important consideration. It is known that both propofol and inhalation agents have a vasodilatory effect in a concentration-dependent manner. However, the extent of reflex tachycardia is quite variable. Compared with the apparent reflex tachycardia with isoflurane, sevoflurane usually does not alter the heart rate. In contrast, propofol inhibits the baroreflex and can even result in bradycardia. In this way, propofol suppresses the cardiac output more than sevoflurane4. The lower intraoperative heart rate might help reduce the amount of intraoperative blood loss.

Few studies have attempted to demonstrate a benefit of a total intravenous anesthesia (TIVA) as the sole technique to optimize and reduce respectively blood pressure levels and bleeding5-9. Besides its potential effects on decreasing peripheral perfusion, other possible benefit of TIVA is the quality of the awakening and the reduced risk of post operative nausea and vomiting (PONV).

Some of the studies on this subject are retrospective in nature with all the biases associated with this type of study. Others, although prospective, measure outcomes based on subjective parameters such as a grading system of the surgeon's appreciation of the difficulty to visualize the operative field due to bleeding, without a correlation with physiologic parameters. Furthermore, not blinding the surgeon to the type of anesthesia may bias the appreciation of the amount of blood loss.

A more objective physiologic measure would be to quantify the blood flow to the mucosa of the sinonasal cavity.

Hypothesis:

Compared to sevoflurane/remifentanyl anesthesia, total intravenous anesthesia with propofol/remifentanyl is associated with lower blood to the sinonasal mucosa, less blood loss and improved surgical field visualization in patients undergoing endoscopic sinus surgery for chronic rhinosinusitis.

Null hypothesis:

Propofol/remifentanyl anesthesia has comparable results to sevoflurane/remifentanyl in terms of blood flow to the sinonasal mucosa, blood loss and surgical field visualization in patients undergoing endoscopic sinus surgery for chronic rhinosinusitis.

Specific Aims Specific Aim 1: Assess nasal blood flow to the sinonasal mucosa using the Rhinolux We will use the Rhinolux system to determine if there are differences in the nasal blood flow between patients with TIVA compared to inhaled anesthesia. The amount of blood flow to the sinonasal mucosa will be measured following induction of general anesthesia with sevoflurane/remifentanyl and compared to the amount of blood flow following induction of general anesthesia with Propofol/remifentanyl. The rhinolux system will be used to measure mucosal blood flow in a continuous fashion until the blood pressure goal is reached. The blood pressure goal will be mean arterial pressure (MAP) of 70, between 60 and 80 mm Hg. A graph with the measurements will be obtained, the time of induction and MAP at goal will be recorded.

The Rhinolux (Rhios GmbH, Germany) is a new non-invasive device that is designed to measure changes in the swelling of the nasal mucosa by a tissue light absorption technique similar to that used in pulse oximetry. The principle is that a light emitter and a detector are placed on two external surface locations opposite each other on the skin, recording the extinction of light that passes the tissue between them as a function of time. The Rhinolux transilluminates the nose at the lower level of the nasal bones, and the light extinction, ∆E measured in optical densities (OD) is proportional to the amount blood in the transilluminated tissue10-12.

Specific Aim 2: Measure the amount of blood loss. Blood loss will be measured by counting the volume in the collection canisters and subtracting the volume of irrigation used intraoperatively. The Neptune Waste Management System (NWMS) will be used for this purpose. The NWMS is a closed suction system that digitally counts the amount of fluid suctioned13. Serum hemoglobin (Hb) will be measured preoperatively in the holding area. Subsequently a 5 mL/kg bolus of normal saline 0.9% or Lactate Ringer will be given within 30 minutes before the start of surgery. Serum Hb will be measured again in the post anesthesia care unit (PACU). Fluid management will be strictly monitored. Maintenance IV fluids will be administered at a rate of 1 ml / kg per hour, including all infusions. Fluid replacement will be performed in a 1 to1 relation with crystalloids (either normal saline 0.9% or Lactate Ringer Solution) for blood loss of less than 5 mL / kg. Colloids will be used for blood loss greater than 5 mL / kg at a volume equal to the blood loss in excess. All fluids given will be recorded in a separate sheet.

Specific Aim 3: Assign a surgical grade score to the operative field. The surgical grade score will be based on the Boezaart surgical risk assessment score, which is a validated and widely accepted score. This is an inexpensive, reliable, and sensitive tool to rapidly evaluate intraoperative bleeding in ESS. The surgical grade score of the operative field will be compared between the groups.

Specific Aim 4: Assess platelet function during anesthesia. To be able to exclude a different explanation for differences in blood loss during surgery, the platelet function will be assessed.

Thromboelastogram- Platelet Mapping. Thromboelastography-Platelet Mapping will be performed on each patient and the results will be compared between the groups. The test will be performed at two different points in time: before induction and in the PACU. This will serve the purpose of determining the baseline platelet function, the effect of the anesthetic combination used and possible changes after surgery has been performed, for each patient.

Thromboelastography is a measure of platelet function15. These test measures blood viscoelastic properties during clot formation. The maximum amplitude in the thromboelastographic trace is dependent on platelet function. Four values that represent clot formation are determined by this test: the R value (or reaction time), the K value, the angle and the MA (maximum amplitude). The R value represents the speed of clot formation (time until the first evidence of a clot is detected). The K value is the time from the end or R until the clot reaches 20 mm and this represents the speed of clot formation. The angle is the tangent of the curve made as the K is reached and offers similar information to K. The MA is a reflection of clot strength. A mathematical formula determined by the manufacturer can be used to determine a Coagulation Index (CI) (or overall assessment of coagulability) which takes into account the relative contribution of each of these 4 values into 1 equation.

In vivo, platelet aggregation tests have indicated in some studies a significant inhibition of platelet function in sevoflurane-anesthetized patients, and after propofol anesthesia, however no change in bleeding time occurred16.

Secondary aim:

Specific Aim 5: Comparison of operative time and quality of recovery. Surgical operating time (SOT) is the time from the moment of injection of local anesthetic in the nasal cavity to the end of application of the local hemostatic agents.

SOT will be documented for each patient and will later be compared between the groups. It is theorized that a decreased blood loss will translate into a shorter operative time.

The quality of recovery will be based on alertness and ventilatory support/oxygenation at arrival in the post anesthesia recovery unit (time from extubation) and 30 minutes after arrival in the PACU, pain control (amount of opioid and non opioid analgesic) at discharge (dismission home after second phase PACU or 23 hours day surgery), abnormal blood pressure or heart rate values to necessitate intervention after PACU transfer, incidence of nausea and vomiting, delay in discharge (if patient in day surgery dismission).

After receiving institutional review board approval and written informed consent, 30 adult patients (ASA I and II) with chronic sinusitis involving a minimum of two paranasal sinuses undergoing ESS will be randomly assigned to receive either sevoflurane/remifentanil (SR) (n=15) or propofol/remifentanil (PR) (n=15) anesthesia. The decision to use 15 patients in each arm is discussed under the statistical analysis section. Patients will undergo the planned endoscopic sinus surgery at Memorial Hermann Hospital-Medical Center and the Ambulatory Care Center at the Memorial Hermann Medical Plaza.

The Lund-MacKay (LM) CT score of the paranasal sinuses will also be obtained. This is a scoring system based on CT scan that categorizes the amount of disease in the sinonasal cavity17 (Table 1). Patients with a total LM score of more than 12 will be defined as high-LM score patients and with a total LM score of 12 or less will be defined as low-LM score patients. In addition at the time of surgery, the surgeon will evaluate and score the amount of edema and redness of the nasal mucosa endoscopically before operation based on the Kupferberg objective endoscopic staging system into stages 0, no evidence of disease; I, edematous mucosa/allergic mucin; II, polypoid mucosa/allergic mucin; and III, polyps and fungal debris18.

A blocked randomization method will be used, to balance patients with regards to the variable of LM score (low or high), It will be important to balance the patients in this aspect since this is a variable that can bias the results.

None of the patients will be pre-medicated. Patients with disease or medication related to coagulation or the cardiovascular system disorders will be excluded. Patients will be blinded to the type of anesthesia administered.

Anesthetic protocol Patients will be premedicated in holding area with dexamethasone and midazolam. The patients will be monitored by American Society of Anesthesia (ASA) standards with ECG, non-invasive blood pressure, pulse oximetry and temperature probe. The blood pressure will be recorded every 2 min for the first 10 minutes then every 5 minutes. Anesthesia will be induced with lidocaine 0.5 mg kg, propofol infusion at 250 mcg/kg/min (to reduce visual bias of propofol infusion) and total volume infused will be adjusted for an induction dose of 2-3 mg/kg before bolus of muscle relaxant, rocuronium 0.5 mg kg in both SR and PR groups. Remifentanil infusion will be started at a rate of 0.4 mcg/kg/min 1-2 minutes before the propofol infusion and a 100 ml 0.9% normal saline bag will be used to blind surgeons in the sevoflurane group. Sevoflurane 1-3% will be administered in group SR, and the infusion of propofol will be stopped. After intubation remifentanil infusion will be changed to 0.2 mcg/kg/min in both groups and propofol will be maintained at 100-150 mcg/kg/min in the TIVA group.

The target mean arterial blood pressure (MAP) will be maintained at 70-80 mm Hg by adjusting the sevoflurane or propofol concentration within their range (between 1-3 vol% for sevoflurane or 100-150 mg ml for propofol) according to the anaesthesiologist's judgement and by surgeon request. If this failed, the remifentanil rate will be adjusted by 0.05 mg kg min. End-tidal CO2 will be continuously monitored (Capnomac Ultima, Datex, Helsinki, Finland) and adjusted to target concentration (Et 32-34 mm Hg) by controlling minute ventilation started from 8 ml kg tidal volume and 10 cycle min respiration rate.

Intravenous fluid administration will be minimized. At induction 5 ml/kg will be used as bolus and a maintenance background infusion of 1 ml/kg/hr will be used in both groups. In order to limit the amount of fluids remifentanil wil be diluted at a concentration of 4 mg in 100 ml.

Postoperative analgesia/PONV. One microgram of fentanyl/kg and/or 0.05 mg of morphine would be given if the patient's numeric rating scale (NRS) of pain is more than 6 before leaving the OR. In the PACU Morphine 1-2 mg IV bolus every 5-10 minutes will be provided as well as ondansetron 4 mg IV bolus. Alternative medications and or supplements will be provided and noted if necessary.

Surgery Protocol

Patients will be positioned in the reverse Trendelenburg and four squeezed cottonoids soaked with a mixed solution of epinephrine and lidocaine (1:100000 epinephrine:lidocaine 2% at 1:1) will be applied topically to each nasal cavity. The surgical procedures will be performed by 3 surgeons with subspecialty training in endoscopic sinus surgery using a similar stepwise technique. The surgeon will not be informed of the type of anesthesia administered. The IV line and solutions will be foiled to prevent the surgeon from seeing the color of the anesthetic agent used.

Statistical analysis

The amount of blood loss and the intraoperative mean remifentanyl infusion rate will be described as the median (1st/3rd quartiles), and will be analyzed using a Mann-Whitney rank sum test. The parameters except for blood loss and the remifentanyl infusion rate will be reported as the mean and standard deviation (SD), and will be analyzed using Student's t-test. The categorical data will be compared using a Chi-square test.

A P-value of .05 will be considered significant. The correlation of the parametric data will be described using the Pearson's correlation coefficients, and the correlation of the non-parametric data will be described using the Spearman's coefficients.

Power analysis: We reviewed studies that compared total intravenous anesthesia to combined anesthesia (inhaled and intravenous) published in the english language through a pubmed search. There were a total of 6 papers available for analysis. The studies found measured different parameters including quantitative and qualitative information. For the purpose of the power analysis we decided to use only the studies measuring blood loss in an objective and quantitive way. The study from Sivaci, et al, had the appropriate information for a power analysis. Thirty two patients were randomly allocated into two different groups. In their study, the average estimated blood loss in the propofol group was 128.1 +/- 37.3 ml compared with an average estimated blood loss of 296.9 +/- 97.8 ml in the sevoflurane group (p<0.01). Their standard deviation was 37.3 and 97.8 respectively. The sample size calculation estimate for an alpha of .05 and a power of 0.8, was of 4 patients in each group. This result is due to the large difference in blood loss between the two groups. However, due to the results from other studies with smaller differences, we decided to use a sample size comparable to what has been used in the literature. Therefore a sample size of 15 was considered appropriate for each arm. We consider that this sample size will have enough patients to detect even a smaller difference than the previously mentioned.

This will be the first study evaluating Rhinolux and regarding this aspect there are no sample size calculations that could be performed.

Estimated sample size for two-sample comparison of means:

Test Ho: m1 = m2, where m1 is the mean in population 1 and m2 is the mean in population 2

Assumptions:

alpha = 0.0500 (two-sided) power = 0.8000 m1 = 128.1 m2 = 296.9 sd1 = 37.3 sd2 = 97.8 n2/n1 = 1.00 Estimated required sample sizes: n1 =4, n2 = 4

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic rhinosinusitis
* Indication by the surgeon of need for endoscopic sinus surgery

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Cattano, MD PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital - Medical Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (16.2) | 50.3 (16) | 50.8 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Volume of Blood Loss
Description: Blood loss was determined by subtracting the volume of irrigation used intraoperatively from the total volume of fluid in the collection canisters.The Neptune Waste Management System will be used for this purpose. This is a closed suction system that digitally counts the amount of fluid suctioned.
Time Frame: during the surgery (from the moment of injection of local anesthetic in the nasal cavity to the end of application of local hemostatis agents, about 1 to 5 hours)
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
milliliters (mL) | 152.9 (161.3) | 355.9 (393.4)

2. Primary Outcome: Number of Participants for Whom Surgical Field Visualization Was Deemed Severely Compromised
Description: Surgeons rated the surgical field using the Boezaart score (which ranges from 0 to 5, with 5 indicating the most compromised surgical field), and this outcome measure reports the number of participants with a Boezaart score of 5. Boezaart scoring is as follows: 0 (No bleeding, cadaveric conditions); 1 (Slight bleeding, no suctioning required), 2 (Slight bleeding, occasional suctioning required; 3 (Slight bleeding, frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed); 4 (Moderate bleeding, frequent suctioning required, and bleeding threatens surgical field directly after suction is removed); 5 (Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible).
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

3. Primary Outcome: Platelet Function as Assessed by Thromboelastography (TEG) Platelet Mapping (PM)
Description: Thromboelastography-Platelet Mapping will be performed to assess the effect of the anesthetics on platelet function. Data are reported as Maximum Amplitude (MA) in millimeters (mm). A greater MA value indicates stronger clotting and greater platelet function.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
millimeters (mm)
  TEG MA [maximum clot strength] | 71.2 (4.80) | 62.3 (11.91)
  adenosine diphosphate channel (ADP) MA [maximum contribution of ADP to clot strength] | 58.2 (10.84) | 42.8 (12.07)
  arachidonic acid channel (AA) MA [maximum contribution of AA to clot strength] | 60.5 (15.01) | 50.6 (14.64)

4. Primary Outcome: Platelet Function as Assessed by Thromboelastography (TEG) Platelet Mapping (PM)
Description: as for outcome 3
Time Frame: During time in post-anesthesia care unit (PACU) (about 30 minutes to 1.5 hours)
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
millimeters (mm)
  TEG MA [maximum clot strength] | 71.9 (5.66) | 68.7 (7.88)
  adenosine diphosphate channel (ADP) MA [maximum contribution of ADP to clot strength] | 51.7 (15.58) | 55.1 (9.20)
  arachidonic acid channel (AA) MA [maximum contribution of AA to clot strength] | 57.7 (19.28) | 57.1 (16.32)

5. Primary Outcome: Nasal Blood Flow to the Sinonasal Mucosa as Assessed by the Rhinolux System
Description: The Rhinolux system was used to measure nasal blood flow (it assessed changes in the swelling of the nasal mucosa by a tissue light absorption technique similar to that used in pulse oximetry)--more negative optical density unit values indicate greater nasal blood flow and less light.
Time Frame: 0-5 minutes after induction of anesthesia
Measure: Mean (Standard Deviation); unit: optical density units
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
optical density units | 0.02 (0.18237) | -0.05 (0.13739)

6. Primary Outcome: Nasal Blood Flow to the Sinonasal Mucosa as Assessed by the Rhinolux System
Description: The Rhinolux system was used to measure nasal blood flow (it assessed changes in the swelling of the nasal mucosa by a tissue light absorption technique similar to that used in pulse oximetry)--negative values indicate greater nasal blood flow and less light.
Time Frame: 60-90 minutes after induction of anesthesia
Measure: Mean (Standard Deviation); unit: optical density units
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
optical density units | -0.11 (0.30615) | -0.41 (0.2583)

7. Secondary Outcome: Duration of Surgery
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
hours | 2.4 (1.2) | 3.6 (1.8)

8. Secondary Outcome: Quality of Recovery as Indicated by Pain Rating Using a Visual Analogue Scale (VAS)
Description: The VAS ranged from 1-10, with 1 being no pain and 10 being worst pain.
Time Frame: During time in post-anesthesia care unit (PACU) (about 30 minutes to 1.5 hours)
Population: These data were not collected for 1 participant in the Inhaled anesthesia arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 10
units on a scale | 3.4 (3.3) | 5.3 (2.8)

9. Secondary Outcome: Quality of Recovery as Indicated by Number of Participants With Nausea
Time Frame: During time in post-anesthesia care unit (PACU) (about 30 minutes to 1.5 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
Participants | 1 | 1

10. Secondary Outcome: Quality of Recovery as Indicated by Recovery Time in the PACU
Time Frame: During time in post-anesthesia care unit (PACU) (about 30 minutes to 1.5 hours)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
minutes | 67 (30.41) | 69 (27.04)

11. Secondary Outcome: Quality of Recovery as Indicated by Number of Participants Who Received an Analgesic Post-operatively
Time Frame: During time in post-anesthesia care unit (PACU) (about 30 minutes to 1.5 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
Number analyzed (Participants) | 12 | 11
Participants
  morphine | 2 | 4
  hydromorphone | 3 | 1
  midazolam | 1 | 1
  meperidine | 2 | 0

ADVERSE EVENTS:
Time Frame: about 2 hours
Arm/Group | Total Intravenous Anesthesia | Inhaled Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes